CLINICAL TRIAL: NCT07118813
Title: Application of Radiomics-based AI Models in Predicting Clinical Outcome of Patients With Renal Cell Carcinoma After Surgical Treatment (AI-Kidney-Prognosis)
Brief Title: Application of Radiomics-based AI Models in Predicting Clinical Outcome of Patients With Renal Cell Carcinoma After Surgical Treatment
Status: Recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0672
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Renal Cell Carcinoma (Kidney Cancer)
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective observational cohort study (AI-Kidney-Prognosis), aiming to non-invasively predict the clinical outcomes in renal cell carcinoma patients after surgical treatment using radiomics-based AI models, thereby assisting clinical decision-making and personalized follow-up strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were treated for renal cell carcinoma in Wuhan Union Hospital from August 2025 to August 2026;
2. Aged > 18 years old;
3. At least one abdominal CT scan before treatment;
4. Tissue biopsy pathological examination confirmed the diagnosis of renal cell carcinoma.

Exclusion Criteria:

1. Poor image quality;
2. Incomplete clinical data or loss of follow-up;
3. Presence of another primary malignancy other than renal cell carcinoma;
4. Unclear pathological diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were treated for renal cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital，Tongji Medical College，Huazhong University of Science and Technology, Wuhan, Hubei, China